CLINICAL TRIAL: NCT03905850
Title: A Randomised, Double-blind, Single Dose, Three Period, Complete Cross Over Trial in Healthy Subjects Investigating the Pharmacokinetics of Subcutaneous Injections of Somapacitan 5 mg/1.5 mL and 10 mg/1.5 mL
Brief Title: A Study to Compare the Uptake Into the Blood of Two Strengths of Somapacitan After Injection Under the Skin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN8640-4491; 2018-003670-27 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1220-5197 (Registry Identifier: World Health Organization (WHO))
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteers; Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somapacitan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Somapacitan 5/10/10 mg (Experimental): One dose of somapacitan 5 mg/1.5 ml followed by two doses of somapacitan 10 mg/1.5 ml. Each dose will be followed by a 3 week observation period.
  Interventions: Drug: somapacitan
- Somapacitan 10/5/10 mg (Experimental): One dose of somapacitan 10 mg/1.5 ml followed by a 5 mg/1.5 ml dose followed by a 10 mg/1.5 ml dose. Each dose will be followed by a 3 week observation period.
  Interventions: Drug: somapacitan
- Somapacitan 10/10/5 mg (Experimental): Two doses of 10 mg/1.5 ml somapacitan followed by a 5 mg/1.5 ml dose. Each dose will be followed by a 3 week observation period.
  Interventions: Drug: somapacitan

INTERVENTIONS:
Drug: somapacitan — 5 mg/1.5 ml and 10 mg/1.5 ml doses administered s.c. (subcutaneously, under the skin)

SUMMARY:
This study will compare two strengths of the new long-acting growth hormone somapacitan. The aim of this study is to test if both strengths are taken up in the blood in the same way. During three separate dosing visits participants will get a total of 3 injections of the study medicine. Somapacitan is not yet approved and therefore cannot be prescribed by a doctor outside of this study. The study duration is between 10 and 15 weeks. Participants will have 17 visits with the study doctor. Three visits will each comprise 6 in-house days with overnight stays. In total, at least 15 overnight stays at the clinic. There will be blood samplings during the study. Participants must come to the clinic regularly for these blood samplings. People who have already received growth hormones in the past or who are growth hormone deficient cannot be in the study. People cannot be in the study if the study doctor thinks that there are risks for their health. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-45 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 18.5 and 24.9 kg/m^2 (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 45 days or 5 times the half-life of the previous investigational medicinal product, whichever is longer, before screening.
* Body weight above 100.0 kg
* Subject with any known history of growth hormone deficiency as declared by the subject.
* Subject who is non-naïve to growth hormone treatment as declared by the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Area under the somapacitan serum concentration time curve from time 0 to the time of the last quantifiable concentration after dosing | 0 to 504 hours after trial product administration
  ng*h/mL
Maximum serum concentration of somapacitan | 0 to 504 hours after trial product administration
  ng/mL

SECONDARY OUTCOMES:
Area under the somapacitan serum concentration time curve from time 0 to 168 hours after dosing | 0 to 168 hours after trial product administration
  ng*h/mL
Area under the somapacitan serum concentration time curve from time 0 to infinity | 0 to 504 hours after trial product administration
  ng*h/mL
Time to maximum serum concentration of somapacitan | 0 to 504 hours after trial product administration
  Hours
Terminal half-life of somapacitan | 0 to 504 hours after trial product administration
  Hours
Area under the insulin-like growth factor I (IGF-I) serum concentration time curve from time 0 to 168 hours after dosing | 0 to 168 hours after trial product administration
  ng*h/mL
Maximum serum concentration of IGF-I after dosing | 0 to 504 hours after trial product administration
  ng/mL
Time to maximum serum concentration of IGF-I after dosing | 0 to 504 hours after trial product administration
  Hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Dombernowsky SL, Damholt BB, Hojby Rasmussen M, Svaerke C, Kildemoes RJ. Investigating the Bioavailability and Insulin-like Growth Factor-I Release of Two Different Strengths of Somapacitan: A Randomised, Double-Blind Crossover Trial. Clin Pharmacokinet. 2024 Jul;63(7):1015-1024. doi: 10.1007/s40262-024-01395-y. Epub 2024 Jul 5. PMID 38969919